CLINICAL TRIAL: NCT03805230
Title: Postoperative Vasopressor Usage : a Prospective International Observational Study (SQUEEZE)
Brief Title: Postoperative Vasopressor Usage: SQUEEZE
Acronym: SQUEEZE
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: SQUEEZE
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Surgical Procedures, Operative; Vasopressor
Keywords: anaesthesia; Intensive Care; vasopressor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: all patients admitted to participating hospitals during 7 consecutive days
- Cohort B: 30 sequential patients with a single additional inclusion criterion

SUMMARY:
A prospective multi-centre international observational study of postoperative vasopressor use, designed to answer the question: 'What is the proportion of patients that receive vasopressor infusions? In the management of these patients;

* Are there variations in the practice between clinicians, hospitals or countries? If yes, are they associated with clinical outcome?
* What are the health economic impacts associated with receiving vasopressors?

DETAILED DESCRIPTION:
Postoperative hypotension is a common occurrence following major non-cardiac surgery and the use of vasopressors in the postoperative period to support blood pressure following optimisation of fluid status is commonplace. Receipt of infused vasopressors postoperatively is considered as a surrogate indicator of significant vasodilation. However, the incidence of postoperative vasopressor therapy has never been described.

By contrast to septic shock, there is no uniform definition of postoperative vasoplegia. Receipt of any amount of vasopressor would provide an objective dichotomous definition but a limitation would be the inability to differentiate degrees of vasodilation. Use of a threshold dose of infused vasopressor to determine a definition is uncomfortably arbitrary. There have been trials of different vasopressors to treat postoperative vasoplegia in cardiac surgical patients and we intend to gather data to inform future design in noncardiac surgery.

In addition, there is evidence of substantial variation in the management of postoperative hypotension between centres, countries and continents. The variation is in assessment (cardiac output and invasive monitoring) and environment (post-operative care units, high-dependency units, ICUs) and management (use and choice of fluids and vasopressors/inotropes). We hypothesise that there is also variation in the incidence of organ dysfunction and the use of organ support, and in clinical outcomes including duration of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery (may be planned or unplanned)
* No plans for return home on the day of surgery, for medical reasons
* Age ≥ 18 on day of surgery

Exclusion Criteria:

* Cardiac surgery
* Obstetric surgery
* Transplant surgery
* Receiving long-term infusions of vasoactive drugs, such as epoprostenol
* Mechanical circulatory support: ventricular assist device, intra-aortic balloon pump, artificial heart or similar
* Already been enrolled in Squeeze

For Cohort B - One additional inclusion criterion:

* Receiving infusion of vasopressors that continues after the patient has left the operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients undergoing any non-cardiac surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of postoperative vasopressor usage in a none cardiac surgical population. | A the primary endpoint is the proportion of patients receiving vasopressor infusions that start between 1 and 24 hours postoperatively
  1. What proportions of patients receive infused vasopressors postoperatively?

CONTACTS AND LOCATIONS:
Overall Officials: Ib Jammer, Dr, Study Chair — Haukeland University Hospital; Ben Creagh-Brown, Study Chair — Royal Surrey County Hospital NHS Foundation Trust
Locations (2):
- University Hospital Knappschaftskrankenhaus Bochum, Bochum, Germany
- Wilhelmina Hospital Assen, Assen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moonesinghe SR, Wong DJN, Farmer L, Shawyer R, Myles PS, Harris SK; SNAP-2 Project team and Steering Group. SNAP-2 EPICCS: the second Sprint National Anaesthesia Project-EPIdemiology of Critical Care after Surgery: protocol for an international observational cohort study. BMJ Open. 2017 Sep 7;7(9):e017690. doi: 10.1136/bmjopen-2017-017690. PMID 28882925
- [Background] Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. Br J Anaesth. 2017 Sep 1;119(3):553. doi: 10.1093/bja/aew472. No abstract available. PMID 28498884
- [Background] Kho ME, Duffett M, Willison DJ, Cook DJ, Brouwers MC. Written informed consent and selection bias in observational studies using medical records: systematic review. BMJ. 2009 Mar 12;338:b866. doi: 10.1136/bmj.b866. PMID 19282440
- [Background] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Lambden S, Creagh-Brown BC, Hunt J, Summers C, Forni LG. Definitions and pathophysiology of vasoplegic shock. Crit Care. 2018 Jul 6;22(1):174. doi: 10.1186/s13054-018-2102-1. PMID 29980217
- [Background] Hajjar LA, Vincent JL, Barbosa Gomes Galas FR, Rhodes A, Landoni G, Osawa EA, Melo RR, Sundin MR, Grande SM, Gaiotto FA, Pomerantzeff PM, Dallan LO, Franco RA, Nakamura RE, Lisboa LA, de Almeida JP, Gerent AM, Souza DH, Gaiane MA, Fukushima JT, Park CL, Zambolim C, Rocha Ferreira GS, Strabelli TM, Fernandes FL, Camara L, Zeferino S, Santos VG, Piccioni MA, Jatene FB, Costa Auler JO Jr, Filho RK. Vasopressin versus Norepinephrine in Patients with Vasoplegic Shock after Cardiac Surgery: The VANCS Randomized Controlled Trial. Anesthesiology. 2017 Jan;126(1):85-93. doi: 10.1097/ALN.0000000000001434. PMID 27841822
- [Background] Abbott TEF, Fowler AJ, Pelosi P, Gama de Abreu M, Moller AM, Canet J, Creagh-Brown B, Mythen M, Gin T, Lalu MM, Futier E, Grocott MP, Schultz MJ, Pearse RM; StEP-COMPAC Group. A systematic review and consensus definitions for standardised end-points in perioperative medicine: pulmonary complications. Br J Anaesth. 2018 May;120(5):1066-1079. doi: 10.1016/j.bja.2018.02.007. Epub 2018 Mar 27. PMID 29661384
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Derived] Jammer I, Martin P, Wunsch H, Debouche S, Harlet P, Moonesinghe R, Forni L, Creagh-Brown B; Writing committee for the Squeeze investigators. Vasopressor use after noncardiac surgery: an international observational study. Br J Anaesth. 2025 Dec;135(6):1609-1617. doi: 10.1016/j.bja.2025.07.034. Epub 2025 Aug 11. PMID 40796492
- [Derived] Creagh-Brown B, Wunsch H, Martin P, Harlet P, Forni L, Moonesinghe SR, Jammer I. The incidence of postoperative vasopressor usage: protocol for a prospective international observational cohort study (SQUEEZE). Perioper Med (Lond). 2023 Mar 24;12(1):8. doi: 10.1186/s13741-023-00296-1. PMID 36964590
- See also: ESAIC Clinical Trial Network website — https://esaic.org/study/squeeze-study/